CLINICAL TRIAL: NCT03477175
Title: An Open-label, Multi-center, Roll-over Study to Assess Long Term Safety of Lenvatinib Monotherapy or Lenvatinib Combination Regimen or Comparator Treatment Arm to Cancer Patients in Eisai Sponsored Lenvatinib Trials
Brief Title: Study to Assess the Long-term Safety of Lenvatinib Monotherapy, a Lenvatinib Combination Regimen, or a Comparator Treatment Arm to Cancer Participants in Eisai Sponsored Lenvatinib Trials
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7080-G000-604; 2017-003668-11 (EudraCT Number)
Record Dates: First submitted 2018-03-20; First posted 2018-03-26 (Actual); Results first posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2023-04

CONDITIONS: Solid Tumors
Keywords: lenvatinib; E7080
MeSH Terms: interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A : Lenvatinib (Experimental): The roll-over eligible participants from Eisai-sponsored lenvatinib studies who received lenvatinib monotherapy or who crossed over from a comparator arm to receive lenvatinib monotherapy in their parent study will continue to receive lenvatinib monotherapy.
  Interventions: Drug: E7080
- Cohort B: Lenvatinib plus Comparator drug (Experimental): The roll-over eligible participants from Eisai-sponsored lenvatinib studies who received lenvatinib combination therapy or who crossed over from a comparator arm to receive lenvatinib combination therapy in their parent study will continue to receive lenvatinib combination therapy.
  Interventions: Drug: E7080; Drug: Comparator Drug
- Cohort C: Comparator drug (Experimental): The roll-over eligible participants from Eisai-sponsored lenvatinib studies who received comparator treatment in their parent study will continue to receive comparator treatment, with exception of participants receiving placebo.
  For China only: The roll-over eligible participants from Eisai-sponsored lenvatinib studies who received comparator treatment in their parent study will continue to receive sorafenib, with exception of participants receiving placebo.
  Interventions: Drug: Comparator Drug; Drug: Comparator Drug: Sorafenib

INTERVENTIONS:
Drug: E7080 — Oral Administration.
  Other Names: lenvatinib; lenvatinib mesilate; lenvatinib mesylate; 4-[3-Chloro-4-(N'-cyclopropylureido)phenoxy]-7-methoxyquinoline-6-carboxamide methanesulfonate
  Arms: Cohort A : Lenvatinib; Cohort B: Lenvatinib plus Comparator drug
Drug: Comparator Drug — Per parent study.
  Arms: Cohort B: Lenvatinib plus Comparator drug; Cohort C: Comparator drug
Drug: Comparator Drug: Sorafenib — Per parent study.
  Arms: Cohort C: Comparator drug

SUMMARY:
This study will be conducted to assess the long-term safety of study drug(s) in participants who are enrolled in Eisai-sponsored lenvatinib studies.

DETAILED DESCRIPTION:
This is an open-label extension study to roll-over eligible participants from Eisai-sponsored lenvatinib studies. The participants may roll-over no sooner than the primary completion dates in their parent study or after all study data for the primary outcome measure have been collected for the parent study. The parent study is defined as the Eisai-sponsored lenvatinib clinical study in which the participant was receiving lenvatinib either as monotherapy or as combination therapy or was receiving any other comparator therapy. The participant can be enrolled in the current study for the purpose of long-term safety data collection if all the selection criteria for the current study are met. The intention is that the participant will not be without study drug during the transition from the parent study to the rollover study.

ELIGIBILITY:
Inclusion Criteria:

It is required for all participants currently participating in other lenvatinib studies to meet the following eligibility criteria.

* Provide signed written informed consent for the roll-over study
* Currently enrolled in an Eisai-sponsored lenvatinib clinical study and still receiving at least one of the study drugs from that protocol
* Currently deriving clinical benefit from at least one of the study drug(s) as determined by the investigator
* Must be able and willing to comply with the current roll-over protocol requirements
* Continued ability to swallow and retain orally administered study drug(s)
* Does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
* Women of childbearing potential and men with reproductive potential (if specified by the parent study) must be willing to continue to use highly effective methods of contraception as per local practices of standard of care during the period of the study
* Women of childbearing potential must have a negative serum pregnancy test at the time of transition to the study and before continuing study drug(s)

Exclusion Criteria:

* Permanent discontinuation of all study drug(s) in the parent study due to toxicity or disease progression and without clinical benefit
* Receiving any prohibited medication(s) as described in the parent study
* Any unresolved toxicity that meets the criteria for study drug(s) discontinuation or withdrawal criteria from the parent study at the time of transition to this study
* Uncontrolled diabetes, hypertension or other medical conditions at the time of transition to the roll-over study that may interfere with assessment of toxicity
* Pregnant or lactating female
* Any serious and/or unstable pre-existing medical condition, psychiatric disorder or other conditions at the time of transition to the roll-over study that could interfere with participant's safety in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (3):
  - Harbor UCLA Medical Center, Torrance, California
  - Northwestern University, Chicago, Illinois
  - Karmanos Cancer Institute, Detroit, Michigan
- The Alfred Hospital, Melbourne, Australia
- Belgium (2):
  - UZ Antwerpen, Edegem, Antwerpen
  - Cliniques Universitaires Saint-Luc, Brussels, Brussels Capital
- China (13):
  - Sun Yat-sen University, Cancer Center, Guangzhou, Guangdong
  - Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Harbin Medical University Cancer Hospital, Haerbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - No.10 People of Shanghai, Shanghai, Shanghai Municipality
  - West China School of Medicine/West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
- Germany (2):
  - Eisai trial site 2, Essen
  - Eisai trial site 1, Würzburg
- Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany, Italy
- Het Nederlands Kanker Instituut Antoni Van Leeuwenhoek Ziekenhuis, Amsterdam, North Holland, Netherlands
- Centrum Onkologii Instytut im.Marii Sklodowskiej Curie-Oddzial w Gliwicach, Gliwice, Poland
- Institutul National de Endocrinologie "C. I. Parhon", Bucharest, Romania
- South Korea (2):
  - National Cancer Center, Goyang-si, Gyeonggido
  - Samsung Medical Center - PPDS, Seoul
- Chulalongkorn University, Pathum Wan, Bangkok, Thailand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 28 investigative sites in China, United States, Australia, Belgium, Germany, Italy, South Korea, Netherlands, Poland, Romania, and Thailand from 16 August 2018 to 21 December 2023.
Pre-assignment Details: A total of 40 participants were screened and enrolled to receive study treatment in this rollover study. The study was to consist of Cohorts A, B and C; however, no participants met criteria for Cohorts B or C, so no participants were enrolled in these cohorts and hence no data were collected and reported for these cohorts. As pre-specified in statistical analysis plan (SAP), data were collected and reported by regions (China and Rest of World) in this study for all sections.
Groups:
- Cohort A, China: Lenvatinib Monotherapy: Participants from China who received lenvatinib monotherapy or who crossed over from a comparator arm to receive lenvatinib monotherapy in their parent study (E7080-C086-108 [NCT03009292], or E7080-C086-308 [NCT02966093]) received lenvatinib dose ranging from 4 milligram (mg) to 24 mg, capsules, orally until progressive disease (PD), unacceptable toxicity, participant's discontinued study, use of nonpermitted concomitant drug, unacceptable noncompliance with the protocol, or lost to follow-up.
- Cohort A, Rest of the World: Lenvatinib Monotherapy: Participants from rest of the world who received lenvatinib monotherapy or who crossed over from a comparator arm to receive lenvatinib monotherapy in their parent study (E7080-E044-101 [NCT00121719], E7080-A001-109 [NCT02686164], E7080-G000-201 [NCT00784303], E7080-G000-303 [NCT01321554], E7080-C086-108 [NCT03009292], or E7080-C086-308 [NCT02966093]) received lenvatinib dose ranging from 4 mg to 24 mg, capsules, orally until PD, unacceptable toxicity, participant's discontinued study, use of nonpermitted concomitant drug, unacceptable noncompliance with the protocol, or lost to follow-up.
Period: Overall Study
Arm/Group | Cohort A, China: Lenvatinib Monotherapy | Cohort A, Rest of the World: Lenvatinib Monotherapy
Started | 19 | 21
Completed | 0 | 0
Not Completed | 19 | 21
Not completed — Unable to travel due to COVID-19 | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Transitioned to commercial drug | 6 | 6
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Adverse Event | 1 | 5
Not completed — Disease Progression | 7 | 7

BASELINE CHARACTERISTICS:
Population: Safety analysis set included the group of participants who received at least 1 dose of study drug.
Groups:
- Cohort A, China: Lenvatinib Monotherapy: Participants from China who received lenvatinib monotherapy or who crossed over from a comparator arm to receive lenvatinib monotherapy in their parent study (E7080-C086-108 [NCT03009292], or E7080-C086-308 [NCT02966093]) received lenvatinib dose ranging from 4 mg to 24 mg, capsules, orally until PD, unacceptable toxicity, participant's discontinued study, use of nonpermitted concomitant drug, unacceptable noncompliance with the protocol, or lost to follow-up.
- Total: Total of all reporting groups
Arm/Group | Cohort A, China: Lenvatinib Monotherapy | Cohort A, Rest of the World: Lenvatinib Monotherapy | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (8.17) | 62.7 (11.45) | 59.6 (10.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 10 | 9 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 21 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 19 | 4 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 17 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Treatment-Emergent Serious Adverse Events (TESAEs)
Description: A treatment-emergent adverse events (TEAE) was defined as an adverse event (AE) that emerged during the treatment in the current roll-over study, having been absent prior to the time the participant signed the current roll-over study informed consent form (ICF), or re-emerged during treatment in the current roll-over study after having been present but resolved before signing the ICF or worsened in severity during treatment in the current roll-over study relative to the pre-ICF state, when the AE was continuous. A serious adverse event (SAE) was any untoward medical occurrence that at any dose: resulted in death; life threatening condition; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect or was medically important due to other reasons than the mentioned criteria.
Time Frame: Up to 58.8 months in current study
Population: Safety analysis set included the group of participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A, China: Lenvatinib Monotherapy | Cohort A, Rest of the World: Lenvatinib Monotherapy
Number analyzed (Participants) | 19 | 21
Participants | 7 | 14

2. Primary Outcome: Number of Participants With Any Non-Serious Treatment-Emergent Adverse Events (TEAEs)
Description: A TEAE was defined as an AE that emerged during the treatment in the current roll-over study, having been absent prior to the time the participant signed the current roll-over study in ICF, or re-emerged during treatment in the current roll-over study after having been present but resolved before signing the ICF or worsened in severity during treatment in the current roll-over study relative to the pre-ICF state, when the AE was continuous. A non-serious TEAE was any AE that was not considered a serious adverse event.
Time Frame: Up to 58.8 months in current study
Population: Safety analysis set included the group of participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A, China: Lenvatinib Monotherapy | Cohort A, Rest of the World: Lenvatinib Monotherapy
Number analyzed (Participants) | 19 | 21
Participants | 18 | 17

3. Primary Outcome: Number of Participants With Treatment-Related TEAEs
Description: A TEAE was defined as an AE that emerged during the treatment in the current roll-over study, having been absent prior to the time the participant signed the current roll-over study ICF, or re-emerged during treatment in the current roll-over study after having been present but resolved before signing the ICF or worsened in severity during treatment in the current roll-over study relative to the pre-ICF state, when the AE was continuous. Related TEAE was defined as AE with causal relationship between the study drug and the TEAE.
Time Frame: Up to 58.8 months in current study
Population: Safety analysis set included the group of participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A, China: Lenvatinib Monotherapy | Cohort A, Rest of the World: Lenvatinib Monotherapy
Number analyzed (Participants) | 19 | 21
Participants | 15 | 14

4. Primary Outcome: Number of Participants With Any TEAE
Description: A TEAE was defined as an AE that emerged during the treatment in the current roll-over study, having been absent prior to the time the participant signed the current roll-over study ICF, or re-emerged during treatment in the current roll-over study after having been present but resolved before signing the ICF or worsened in severity during treatment in the current roll-over study relative to the pre-ICF state, when the AE was continuous.
Time Frame: Up to 58.8 months in current study
Population: Safety analysis set included the group of participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A, China: Lenvatinib Monotherapy | Cohort A, Rest of the World: Lenvatinib Monotherapy
Number analyzed (Participants) | 19 | 21
Participants | 18 | 20

ADVERSE EVENTS:
Time Frame: Up to 58.8 months in current study
Description: Safety analysis set included the group of participants who received at least 1 dose of study drug.
Arm/Group | Cohort A, China: Lenvatinib Monotherapy | Cohort A, Rest of the World: Lenvatinib Monotherapy
All-Cause Mortality (participants affected / at risk) | 2/19 | 5/21
Serious Adverse Events (participants affected / at risk) | 7/19 | 14/21
Other Adverse Events (participants affected / at risk) | 18/19 | 17/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A, China: Lenvatinib Monotherapy (N=19) | Cohort A, Rest of the World: Lenvatinib Monotherapy (N=21)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A, China: Lenvatinib Monotherapy (N=19) | Cohort A, Rest of the World: Lenvatinib Monotherapy (N=21)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (17) | 4 (11)
Gingival disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 1 (2) | 1 (2)
Peripheral swelling (General disorders) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 4 (4) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (5)
Alanine aminotransferase increased (Investigations) | 4 (5) | 1 (1)
Albumin globulin ratio decreased (Investigations) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 1 (2) | 0 (0)
Apolipoprotein A-I decreased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (7) | 1 (1)
Bile acids increased (Investigations) | 1 (3) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 2 (3) | 1 (1)
Blood bicarbonate decreased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 2 (5) | 1 (3)
Blood fibrinogen decreased (Investigations) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (7) | 1 (2)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (2) | 0 (0)
Low density lipoprotein increased (Investigations) | 1 (4) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0)
Platelet count increased (Investigations) | 1 (1) | 0 (0)
Platelet-large cell ratio decreased (Investigations) | 1 (1) | 0 (0)
Protein total decreased (Investigations) | 1 (2) | 0 (0)
Urinary occult blood positive (Investigations) | 2 (4) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 5 (9)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 (6) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 (9) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (5)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (4)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Albuminuria (Renal and urinary disorders) | 4 (13) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 3 (4)
Proteinuria (Renal and urinary disorders) | 6 (13) | 1 (5)
Renal failure (Renal and urinary disorders) | 1 (3) | 0 (0)
Vulvovaginal inflammation (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (3) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT03477175/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-28): https://cdn.clinicaltrials.gov/large-docs/75/NCT03477175/SAP_001.pdf